CLINICAL TRIAL: NCT05523622
Title: Comparison of Intraocular Pressure Measurement With the Novel TonoVera Device With Other Commonly Used Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Reichert, Inc. (Industry)
Responsible Party: Principal Investigator, Catherine Seeger, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UB Tono-Vera Comparison Trial
Record Dates: First submitted 2022-08-22; First posted 2022-08-31 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: We are comparing the accuracy of eye pressure measurements with a Tono-Vera device compared to the current gold standard, Goldmann Applanation Tonometry.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- IOP Measurement (Other): These are the measurements of the intraocular pressure.
  Interventions: Device: Tono-Vera tonometer; Device: Goldman Applanation Tonometry

INTERVENTIONS:
Device: Tono-Vera tonometer — The tonometer measures intraocular pressure with a small rebound probe, similar to those used with other tonometers currently on the market, such as the iCare.
Device: Goldman Applanation Tonometry — This is the current gold standard for measuring eye pressure.

SUMMARY:
We are testing the accuracy of Reichert's Tono-Vera tonometer by comparing measurements of IOP with this device and measurements with other commonly-used tonometers, including Goldmann Applanation and iCare.

DETAILED DESCRIPTION:
This is a comparative study between the TonoVera, the gold standard Goldmann Applanation Tonometry (GAT) and an established rebound tonometry device, iCare. IOP measurements will be obtained using the following devices: Reichert's prototype Tono-Vera Rebound tonometer (a rebound tonometer in development), iCare's iC100 rebound tonometer (a device commonly used in clinical practice), GAT (a device commonly used in clinical practice). Reichert's iPac Handheld Pachymeter (a device commonly used in clinical practice) will be used to measure the test subject's Central Corneal Thickness (CCT), measured in µm if CCT is not already on file. An Autorefractor Keratometer (ARK) (a device commonly used in clinical practice) will be used to measure necessary vision correction and corneal curvature. The Ocular Response Analyzer (a device commonly used in clinical practice) will be used to measure corneal hysteresis. Multiple IOP measurements will be taken with each device on each eye for all subjects: 3 along the central cornea, 3 along the peripheral cornea, and 3 along the sclera.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide signed and dated informed consent form. Patients willing to comply with all study procedures and be available for the duration of the study.

Male or female patients aged 18 to 99 Patients in good general health as evidenced by ability to come to their appointment on day of study.

Exclusion Criteria:

* Patients age less than 18 years Patients unable or unwilling to provide informed consent to participate in the study Patients for which an accurate tonometry reading cannot be performed. This may include those with blepharospasm (lid squeezers), nystagmus, extensive corneal pathology, or contact lens wearers who cannot remove their contact lens.Patients with significant scleral thinning Patients with a known allergy to proparacaine or fluorescein as these are used to anesthetize and allow measurement respectively of the eye when used with the Goldmann tonometer.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure | Baseline only
  pressure inside the eye

CONTACTS AND LOCATIONS:
Locations (1):
- Ross Eye Institute, Buffalo, New York, United States

REFERENCES:
- [Background] Chen M, Zhang L, Xu J, Chen X, Gu Y, Ren Y, Wang K. Comparability of three intraocular pressure measurement: iCare pro rebound, non-contact and Goldmann applanation tonometry in different IOP group. BMC Ophthalmol. 2019 Nov 14;19(1):225. doi: 10.1186/s12886-019-1236-5. PMID 31726999
- [Background] Hager A, Loge K, Schroeder B, Fullhas MO, Wiegand W. Effect of central corneal thickness and corneal hysteresis on tonometry as measured by dynamic contour tonometry, ocular response analyzer, and Goldmann tonometry in glaucomatous eyes. J Glaucoma. 2008 Aug;17(5):361-5. doi: 10.1097/IJG.0b013e31815c3ad3. PMID 18703945
- [Background] Kaushik S, Pandav SS, Banger A, Aggarwal K, Gupta A. Relationship between corneal biomechanical properties, central corneal thickness, and intraocular pressure across the spectrum of glaucoma. Am J Ophthalmol. 2012 May;153(5):840-849.e2. doi: 10.1016/j.ajo.2011.10.032. Epub 2012 Feb 4. PMID 22310080